CLINICAL TRIAL: NCT06695065
Title: Value of Speckle Tracking Echocardiography in Early Assessment of Cardiac Function in Inflammatory Bowel Disease Patients
Brief Title: Value of Speckle Tracking Echocardiography Inflammatory Bowel Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa AbdelShafy mohamed, Physician, Assiut University
Other Study IDs: Echocardiogray in IBD
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-11

CONDITIONS: Echocardiography; Inflammatory Bowel Diseases; Cardiac Function
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Study group adult with ulcerative colitis: 50 Adult patients with ulcerative colitis
- control group: 50 age and sex matched control group.

SUMMARY:
Value of speckle tracking echocardiography in early assessment of cardiac function in inflammatory bowel disease .

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a common form of inflammatory bowel disease (IBD) that consists of chronic inflammatory disorders of the colon and the small intestine with unknown etiology. Chronic inflammation is the basis of complicated pathogenesis, and the course of the disease is often complicated by an immune response. Malnutrition, malabsorption and the involvement of organs other than those of the gastrointestinal tract are frequent consequences of the disease . Although extra-intestinal manifestations of IBD are common (ranging from 6% to 47%), cardiac involvement is rare.

Inflammatory bowel disease (IBD) is a known risk factor for cardiovascular disease (CVD). IBD patients have a two- to threefold increased risk of venous thromboembolism, particularly during acute flares when disrupted homeostasis of anti- and procoagulants leads to a hypofibrinolytic state. Cardiovascular manifestations in Crohn's disease (CD) and ulcerative colitis (UC) include conditions such as Takayasu's arteritis, pericarditis, and myocarditis. Chronic inflammation and altered lipid metabolism, along with long-term use of anti-inflammatory drugs (e.g., corticosteroids, TNF-α inhibitors), are thought to drive CV pathology in IBD. Additionally, chronic inflammation is linked to pathological collagen deposition in affected organs.

Although conventional echocardiography is a widely accessible and easy tool to detect cardiac abnormalities, novel echocardiographic techniques and indices offer easy, reproducible and quantitative information for evaluating left ventricle function and subclinical changes . Speckle tracking echocardiography (STE) is an advanced echocardiographic methodology for the quantification of myocardial function. STE has been successfully used to identify early subclinical cardiac involvement in a variety of asymptomatic populations with chronic diseases and unremarkable conventional echocardiography. Unlike earlier echocardiography techniques, two-dimensional speckle tracking echocardiography (2DSTE) is less angle-dependent. In addition, STE is not affected by the rotation of the heart and allows heart functions to be examined segment by segment from various echocardiographic views . Despite, studies have examined subclinical cardiac impairment in patients with IBD, to the best of our knowledge, none have explored the impact of ulcerative colitis activity on cardiac function through using STE.

ELIGIBILITY:
Inclusion Criteria:

* Age (18-60) yrs.
* Both sexes.
* Patients with IBD either in active form or in remission.

Exclusion Criteria:

* Patients with ischemic heart disease. -Patients with other comorbidities affecting heart as uncontrolled hypertension or diabetes. -
* Pregnant females.
* Malignancy

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: History:
  Demographic data; age, sex. History of the disease: onset, duration, medication. Family history of disease. History of comorbidities: hypertension, diabetes, ischemic heart diseases.
  Laboratory investigations:
  Fasting blood glucose, 2 hr postprandial and glycated haemoglobin A1c (HbA1c). Lipid profile: LDL, HDL, triglyceride, cholesterol. Inflammatory markers: CRP, ESR Complete blood picture Evaluation of Disease Severity Partial Mayo score consists three of the four components of the standard Mayo score, excluding endoscopic findings (stool frequency, rectal bleeding and physician's global assessment). Each component is assigned a score of 0-3, and total score ranges from 0 to 9 for each patient.
  -Echocardiographic Examination
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Subclincal cardiovascular events in IBD patients. | through study completion, an average of 2 year
  Assessment the predictive ability of Speckle TRACKING Echocardiograpy in development of subclinical cardiovascular events in IBD patients.
Relation between isease activity and cardiac function | through study completion, an average of 2 year
  Evaluation of the relationship between disease activity and cardiac function as measured by Speckle tracking Echocardiograpy.

SECONDARY OUTCOMES:
correlation of Speckle TRACKING Echocardiograpy findings with traditional echocardiographic parameters | through study completion, an average of 1 year
  Detection of correlation of Speckle TRACKING Echocardiograpy findings with traditional echocardiographic parameters and inflammatory markers.